CLINICAL TRIAL: NCT01835860
Title: Prostatic Artery Embolization for Benign Prostatic Hyperplasia
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Saskatchewan Health Authority - Regina Area (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REB-12-81
Record Dates: First submitted 2013-03-27; First posted 2013-04-19 (Estimated); Last update posted 2016-04-07 (Estimated); Status verified 2016-04

CONDITIONS: Benign Prostate Hyperplasia
Keywords: BPH
MeSH Terms: conditions — Prostatic Hyperplasia

ARMS (1):
- Embolization (Other): Prostate artery embolization
  Interventions: Procedure: Prostate artery embolization

INTERVENTIONS:
Procedure: Prostate artery embolization

SUMMARY:
To evaluate whether Prostatic Artery Embolization (PAE) might be an effective alternative treatment option for benign prostatic hyperplasia (BPH), in comparison to current gold standard surgical treatment- Transurethral Resection of Prostate (TURP).

ELIGIBILITY:
Inclusion Criteria:

1. Moderate to severe lower urinary tract symptoms (i.e. International prostate symptom score IPSS>8) who are bothered by their symptoms (i.e., interfere with the daily activities of living)
2. Urinary retention (related to BPH) leading to catheterization.
3. Refractory to medical treatment or patient is not willing to consider medical treatment
4. Pre trans-urethral resection of prostate (TURP) to reduce the size of prostate gland if prostate is too big for TURP surgery.

Exclusion Criteria:

1. Mild symptoms (IPSS <8)
2. Moderate to severe lower urinary tract symptoms (i.e. IPSS>8) who are not bothered by their symptoms (i.e., symptoms do not interfere with the daily activities of living).
3. Suspected malignancy.
4. Any of the following clearly related to BPH- bladder stones, recurrent UTIs, and renal insufficiency.
5. Advanced atherosclerosis and unsuitable vascular access.
6. Allergy to intravenous contra

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2013-03; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline in symptom severity at 1, 3, 6 and 12 months follow-up, as measured by International prostate symptoms score (IPSS). | 1, 3, 6 and 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Regina General Hospital, Regina, Saskatchewan, Canada